CLINICAL TRIAL: NCT06898398
Title: Transcatheter Arterial Chemoembolization Combined Surgery Versus Surgery for the Resectable Huge Hepatocellular Carcinoma: a Multicenter Propensity Analysis
Brief Title: TACE Combined Surgery for the Resectable Huge HCC
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhou Qunfang, Clinical Professor, Sun Yat-sen University
Other Study IDs: Liver Project 15
Record Dates: First submitted 2025-03-21; First posted 2025-03-27 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Hepatocellular Carcinoma; Hepatic Chemotherapy; Liver Cancer; Surgery
Keywords: huge hepatocellular carcinoma; TACE; Surgery
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TACE+surgery: patients underwent neoadjuvant TACE followed by surgical treatment.
  Interventions: Procedure: TACE; Procedure: Surgery
- Surgery: patients underwent surgical treatment.
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: TACE — TACE procedure was a 2.8-F microcatheter was super-selectively inserted into the tumor feeding artery using the coaxial technique. Then a combination of lipiodol (5-15 ml), lobaplatin (30-50 mg), and Pirarubicin (30-50 mg) was infused into each tumor. We defined technical success as complete embolization of the tumor-feeding artery resulting in no tumor staining observed by angiogram at the end of procedure.
  Groups: TACE+surgery
Procedure: Surgery — The surgical plan was based on the tumor size, tumor location, and liver function. We applied Pringle's maneuver with cycles of clamping and unclamping times of 1-10 and 5 min, respectively, and maintained the central venous pressure below 4 mmHg during parenchymal dissection to control intraoperative bleeding.

SUMMARY:
Huge hepatocellular carcinoma (HCC) is defined as a tumor with a maximum diameter greater than 10 cm. With advancements in surgical techniques, hepatectomy can be performed safely in some patients with huge HCC without vascular invasion or distant metastasis and with preserved liver function. The high risk of recurrence after surgery is another challenge for surgeons. Neoadjuvant TACE has been shown to improve the clinical outcomes of patients with HCC, especially those with a high risk of recurrence, such as those with multinodular tumors, large tumors, and tumor thrombus. The present multicenter study aimed to evaluate the efficacy of neoadjuvant TACE in patients with huge HCC who underwent liver resection.

DETAILED DESCRIPTION:
Huge hepatocellular carcinoma (HCC) is defined as a tumor with a maximum diameter greater than 10 cm. With advancements in surgical techniques, hepatectomy can be performed safely in some patients with huge HCC without vascular invasion or distant metastasis and with preserved liver function. However, the 2-year recurrence rate in such cases is as high as 70%, indicating the need for more effective interventions to improve outcomes. Neoadjuvant TACE has been shown to improve the clinical outcomes of patients with HCC, especially those with a high risk of recurrence, such as those with multinodular tumors, large tumors, and tumor thrombus. The impact of neoadjuvant TACE on the long-term oncological outcomes of huge HCC requires investigation. The present multicenter study aimed to evaluate the efficacy of neoadjuvant TACE in patients with huge HCC who underwent liver resection.

ELIGIBILITY:
Inclusion Criteria:

1. clinical or pathological diagnosis of primary HCC;
2. tumor diameter > 10 cm on images before inclusion;
3. age 18 to 75 years;
4. no macrovascular invasion or extrahepatic metastasis;
5. liver resection with complete removal of the tumor and adequate remnant liver volume;
6. albumin-bilirubin (ALBI) grade I and II;
7. Eastern Cooperative Oncology Group performance status (ECOG) score of 0-1;
8. hemoglobin level ≥ 8.5 g/dL, total bilirubin level ≤ 30 mmol/L, alanine transaminase (ALT) and aspartate aminotransferase (AST) levels ≤ 5 × upper limit of normal, serum creatinine level ≤ 1.5 × upper limit of normal;
9. prothrombin time ≤ 18 s or international normalized ratio < 1.7.

Exclusion Criteria:

1. HCC with macrovascular invasion or extrahepatic metastasis;
2. tumor with a maximum diameter ≤ 10 cm on images before inclusion;
3. recurrent HCC;
4. serious medical comorbidities;
5. portal hypertension, including presence of either esophageal varices or splenomegaly with a platelet count less than 109/L;
6. cardiac ventricular arrhythmias requiring anti-arrhythmic therapy;
7. incomplete data or lost to follow-up within three months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is a multicenter, observational real-world study to compare the efficacy of TACE with surgery inhuge hepatocellular carcinoma. This study focused on the management of locoregional therapy combined surgery. This study will create a database that will provide clinical parameters and outcomes of patients undergoing combined therapy for huge HCC therapy.
Sampling Method: Probability Sample
Enrollment: 326 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival （RFS） | 24 months
  RFS was defined as the time from surgery to tumor progression or the last follow-up

SECONDARY OUTCOMES:
Overall survival (OS) | 60 months
  OS was defined as the time from surgery to death or the last follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Feng Duan, MD, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA general hospital, Beijing, Beijing Municipality, China